CLINICAL TRIAL: NCT01098552
Title: Participation in Procurement of Tissue, Serum, Plasma, Cell Bank, DNA and RNA Samples, and Urine for Biological Studies Related to Prostate Cancer and Prostate Cancer Treatment Follow Up
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Robert Karnes, Principal Manager, Mayo Clinic
Other Study IDs: 1937-00; Mayo Clinic Prostate SPORE
Record Dates: First submitted 2010-04-01; First posted 2010-04-02 (Estimated); Last update posted 2013-01-11 (Estimated); Status verified 2013-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, prostate tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- High-risk radical prostatectomy patients
- Primary external beam radiotherapy patients
- Primary prostate brachytherapy patients
- Hormone refractory prostate cancer patients
- Active Surveillance
- Prostate biopsy patients

SUMMARY:
This research study is being done to collect regular and routine follow-up information related to the outcome of treatment for prostate cancer.

This study is also being done to relate treatment outcome to measurement of substances in the blood such as prostate-specific antigen (PSA) and other markers. Also environmental and genetic factors that might be responsible for prostate cancer are being investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent explained and signed prior to any study related procedures.
2. Age ≥18 years
3. Eastern Cooperative Oncology Group (ECOG) performance status of 2 or better, or Karnofsky performance of 60% or better.
4. Histologically confirmed adenocarcinoma of the prostate within 10 years of study entry.
5. Willingness to return to Mayo Clinic Rochester for follow-up or participate in mail-in PSA processing.
6. Must be disease-free from a previous diagnosis of cancer for a period of time = 5 years excluding cutaneous malignancies of squamous cell or basal cell carcinoma.

Exclusion Criteria:

1. Life expectancy < 5 years.
2. Inability to return to Mayo Rochester for follow-up appointments, sera, and urine collection per protocol.
3. Previous or a concurrent diagnosis of cancers other than basal cell or invasive squamous cell carcinoma of skin within the past 5 years.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There are six patient cohorts which are being recruited to the Prostate Clinical Follow-up Core in support of the Specialized Program of Research Excellence (SPORE). The six groups are: 1. High-risk radical prostatectomy patients, 2. Primary external beam radiotherapy patients, 3. Primary prostate brachytherapy patients, 4. Hormone refractory prostate cancer patients, 5. Active Surveillance. 6. Prostate biopsy patients. The inclusion criterion for group 6 is that the patient is scheduled to undergo a prostate biopsy for the purposes of definitive prostate cancer diagnosis. There are no exclusion criteria for group 6.
Sampling Method: Non-Probability Sample
Enrollment: 4900 (Actual)
Dates: Start 2010-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R. J. Karnes, MD, Study Director — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States